CLINICAL TRIAL: NCT01922752
Title: An Open-Label Study to Determine the Maximum Tolerated Dose of Oral CEP-37440 Administered as a Single Agent in Patients With Advanced or Metastatic Solid Tumors
Brief Title: To Determine the Maximum Tolerated Dose of Oral CEP-37440 in Patients With Advanced or Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C37440/1108
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Last update posted 2021-11-12 (Actual); Status verified 2021-11

CONDITIONS: Solid Tumors
Keywords: CEP-37440; Advanced solid tumors; Metastatic solid tumors
MeSH Terms: interventions — CEP-37440

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CEP-37440 (Experimental)
  Interventions: Drug: CEP-37440

INTERVENTIONS:
Drug: CEP-37440 — CEP-37440 will be supplied as 25 mg and 100 mg capsules and will be orally administrated daily.
  Patients will be enrolled sequentially in dose escalating cohorts to receive CEP-37440 until a maximum tolerated dose has been defined.

SUMMARY:
The primary objective is to determine the maximum tolerated dose (MTD), safety, and tolerability of oral CEP-37440 administered daily to patients with advanced or metastatic solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologic or cytologic evidence of a solid neoplasm for which no standard therapy is available, or have progressed despite standard therapy, or are intolerant to standard therapy.
* Patients must have evidence of recurrent, locally advanced, or metastatic disease.
* Patients can either have had no prior anticancer therapy, multiple lines of either prior chemotherapy/biologic therapy/experimental therapy or, if the patient has anaplastic lymphoma kinase (ALK)-positive non-small cell lung cancer (NSCLC), prior crizotinib.
* Patients must have a predicted life expectancy of more than 3 months.
* Patients must have presence of at least 1 lesion that is measurable or evaluable using RECIST v1.1.
* Patients must have an ECOG performance score of 0, 1, or 2.
* Patients with central nervous system (CNS) metastases will be allowed on this study. Patients may have received surgical and/or radiation treatment. The metastases must be neurologically stable, on or off corticosteroids. Patients can have low level, asymptomatic brain lesions that do not require surgical/radiation intervention acutely. Patients with symptomatic lesions with impending neurologic compromise should be appropriately treated with high dose steroids/radiation and may be re-evaluated for this study when neurologically stable.
* Patients must have completed any prior anticancer treatment and must have recovered from any acute toxicities. The period between the last dose of prior treatment and the first dose of study drug treatment must be at least 1 week for radiotherapy and at least 2 to 3 weeks for all other modalities of therapy including chemotherapy, monoclonal antibody therapy, immunotherapy, other investigational drugs, or other kinase inhibitors.
* Other criteria apply.

Exclusion Criteria:

* The patient has ongoing or active infection requiring parenteral antibiotics.
* The patient has uncontrolled hypertension despite adequate therapy (ie, systolic blood pressure higher than 150 mm Hg or diastolic blood pressure higher than 90 mm Hg found on 2 separate occasions separated by 1 week).
* The patient has uncontrolled diabetes mellitus (despite therapeutic intervention) and occurrence of more than 2 episodes of ketoacidosis in the 12 months prior to the first dose of study drug.
* The patient has an active second malignancy other than curatively resected basal cell carcinoma of the skin, squamous cell carcinoma of the skin, in situ carcinoma of the cervix, or other cancers for which they are treated with curative intent, and no known active disease in the 3 years prior to enrollment.
* The patient has a primary brain tumor. Patients may have brain metastases from another primary site.
* The patient has QTcF interval greater than 450 msec, has a known history of QTcF prolongation, is taking medications known to prolong QTcF, or has a history of torsade de pointes.
* The patient has a prior ALK-inhibitor-related toxicity or any other prior therapy-related acute toxicity that has not resolved prior to the first dose of study drug.
* Other criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors (RECIST v1.1) | 8 months

SECONDARY OUTCOMES:
Time to Response (TTR) | 8 months
  The time interval from the date of first dose to the first documented response (complete or partial response)
Number of participants with adverse events | From signing of the informed consent to the end of the follow-up visit (approximately Month 10)
Time to Progression (TTP) | 8 months
  The time interval from date of first dose to first documented disease progression
Progression-free Survival (PFS) | 10 months
  Time interval from date of first does to first documented disease progression or death from any cause (whichever occurs first)
Time to New Metastases (TTNM) | 8 months
  Time interval from date of first dose to first documented new metastatic lesion not reported at baseline

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Teva Investigational Site 10689, Chicago, Illinois
  - Teva Investigational Site 10687, Philadelphia, Pennsylvania
  - Teva Investigational Site 10686, San Antonio, Texas

REFERENCES:
- [Derived] Schilder RJ, Rasco D, Sharma MR. An open-label study to determine the maximum tolerated dose of oral ESK-440 administered as a single agent in patients with advanced or metastatic solid tumors. Neoplasia. 2025 Mar;61:101133. doi: 10.1016/j.neo.2025.101133. Epub 2025 Feb 5. PMID 39914170